CLINICAL TRIAL: NCT06026020
Title: Exploration of the Pathogenesis of Intestinal Behcet's Syndrome: a Single-center Prospective Observational Study
Brief Title: Pathogenesis of Intestinal Behcet's Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K4434
Record Dates: First submitted 2023-08-17; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Behcet's Syndrome, Intestinal Type
Keywords: Behcet's syndrome; intestinal Behcet's syndrome; inflammatory bowel disease; microbiome; metabolomics
MeSH Terms: conditions — Behcet Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Behcet's syndrome patients with intestinal involvement
  Interventions: Other: Biological samples collection
- Behcet's syndrome patients without intestinal involvement
  Interventions: Other: Biological samples collection
- Inflammatory bowel disease patients
  Interventions: Other: Biological samples collection
- Health control
  Interventions: Other: Biological samples collection

INTERVENTIONS:
Other: Biological samples collection — Samples of blood, faeces, saliva are collected for analysis.

SUMMARY:
There is a direct interaction between food, intestinal flora and the intestinal barrier composed of intestinal epithelial cells and mucosal immunity, whose composition and functional alterations are theorized to be closely related to the development of gastrointestinal (GI) involvement in Behcet's syndrome (BS) patients. Therefore, this study focuses on the population of patients with intestinal BS and explores the unique mechanisms leading to intestinal involvement in BS patients in terms of the characteristics of intestinal microecology. Since oral ulcers are one of the most common clinical manifestations in BS patients, in addition to intestinal flora analysis, this application project also plans to collect saliva samples from patients in the hope of obtaining a holistic understanding of mucosal flora in different parts of the entire GI tract. Serological testing and analysis will also be performed, focusing on changes in the intestinal tract and serum IgE levels, and analyzed in conjunction with microbiomics to provide evidence to further elucidate the pathogenesis of BS and GI involvement, and to search for more efficient therapeutic strategies, in terms of a variety of aspects, including clinical manifestations and disease progression.

ELIGIBILITY:
Inclusion Criteria:

Behcet's syndrome patients with intestinal involvement:

* Attendance at Peking Union Medical College Hospital, fulfillment of one of the two diagnostic criteria for BS (1990 Criteria of International Study Group for Behcet's disease or 2014 International Criteria for Behçet's Disease), and well-documented medical records;
* Age 20-65 years old;
* Have evidence of GI involvement, including clinical manifestations, laboratory tests, endoscopy, imaging and pathology;
* Signed written informed consent and willingness to cooperate.

Behcet's syndrome patients with intestinal involvement:

* Attendance at Peking Union Medical College Hospital, fulfillment of one of the two diagnostic criteria for BS (1990 Criteria of International Study Group for Behcet's disease or 2014 International Criteria for Behçet's Disease), and well-documented medical records;
* Age 20-65 years old;
* Have no evidence of GI involvement, including clinical manifestations, laboratory tests, endoscopy, imaging and pathology;
* Signed written informed consent and willingness to cooperate.

Inflammatory bowel disease patients:

* Attended Peking Union Medical College Hospital and was diagnosed with Crohn's disease by a combination of clinical, imaging, and pathologic diagnosis;
* Age 20-65 years old;
* Signed written informed consent and willingness to cooperate.

Health controls:

* Healthy individuals aged 20-65 years;
* Signed written informed consent and willingness to cooperate.

Exclusion Criteria:

* Other systemic diseases, such as autoimmune diseases, infectious diseases, malignant tumors, etc;
* Patients with other intestinal diseases, such as intestinal tumors, intestinal tuberculosis, intestinal infections;
* Patients with other oral diseases, such as cavity caries, oral abscesses, oral tumors, oral candidiasis, and dry mouth;
* Patients taking antibiotics and probiotics within one month.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient who have Behcet's syndrome with or without intestinal involvement, compared with inflammatory bowel disease patients and health controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Structure and composition of gut microbiota | Day 1 after addmission due to the disease activity and signing an informed consent (for patients); or day 1 after signing an informed consent (for health controls)
  DNA extraction from stool samples will be tested through 16S microbial sequencing and metagenomic sequencing to establish and compare microbial profiles of the gut microbiota among different groups.
Structure and composition of oral microbiota | Day 1 after addmission due to the disease activity and signing an informed consent (for patients); or day 1 after signing an informed consent (for health controls)
  DNA extraction from saliva samples will be tested through 16S microbial sequencing and metagenomic sequencing to establish and compare microbial profiles of the oral microbiota among different groups.
Structure and composition of metabolomics | Day 1 after addmission due to the disease activity and signing an informed consent (for patients); or day 1 after signing an informed consent (for health controls)
  Serum extraction from blood samples will be tested through non-targeted metabolomics techniques to analysis and compare metabolomics among different groups.
Serum level of Immunoglobulin E | Day 1 after addmission due to the disease activity and signing an informed consent (for patients); or day 1 after signing an informed consent (for health controls)
  Serum extraction from blood samples will be used to test and compare the level of IgE among different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No